CLINICAL TRIAL: NCT06097494
Title: Healthcare Disparities in Vitiligo: a Population-based Cohort Study in the UK
Brief Title: Investigating Healthcare Disparities in Vitiligo
Status: Completed | Type: Observational
Sponsor: Momentum Data (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: P084
Record Dates: First submitted 2023-10-09; First posted 2023-10-24 (Actual); Results first posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2024-10

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- People with Vitiligo: Children and adults with new onset Vitiligo registered with OPCRD during the study period.
  Interventions: Other: No intervention
- People without Vitiligo: Children and adults without Vitiligo registered with OPCRD during the study period
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Observational analysis of usual care only.

SUMMARY:
Vitiligo is an acquired, non contagious skin disorder characterised by depigmented patches of skin that may appear in a localised or very generalised distribution, and affecting 0.5-2.0% of the global population.There are however, limited population-based studies on the burden of vitiligo and disparities across people of different ethnicities and deprivation.

The overall purpose of this study is to provide an estimate of the lifetime risk of vitiligo in the population overall and by sociodemographic subgroups. Moreover, to do a subgroup analysis in the vitiligo population to identify health-related disparities across people in different sex, age, deprivation and ethnicity. A detailed understanding of the burden of disease in different sociodemographic groups is vital to plan resource provision.

DETAILED DESCRIPTION:
This study will provide estimate of the cumulative lifetime risk of vitiligo in the population overall, and by important sociodemographic groups, including age, sex, ethnicity and deprivation, which will prevalent key data to show the relative burden of vitiligo across the aforementioned groups. These approaches allow creation of cumulative lifetime risk plots which provide an excellent and accessible way to display the relative disease burden across groups.

The cumulative lifetime risk of vitiligo will be estimated at age 80 years (approximate lifetime expectancy in the UK) using survival models, with age as the timescale and accounting for competing risk of death.

This study will also perform a subgroup analysis in the vitiligo population to identify health-related disparities across people in different deprivation, sex and ethnic groups. The disparities that will be considered are: Mental health conditions; healthcare utilisation; and work impact (time off work and unemployment),

The assessment of any associations with baseline characteristics and the outcome of interest will be used using Cox proportional hazards models (time to event outcomes) and generalised linear models.

ELIGIBILITY:
Inclusion Criteria:

* The cohort for the endpoint analysis will consist of all adults and adolescents (aged 13+) contributing to OPCRD during the study period (2004-2020).
* The cohort for the lifetime risk analysis will consist of all people contributing to OPCRD during the study period.
* The vitiligo cohort consists of people newly diagnosed with vitiligo at any point during the study period.

Exclusion Criteria:

* People with the alternative non-vitiligo diagnoses (other hypopigmenting conditions).
* People with vitiligo diagnosis within 6 months of practice registration.
* People without vitiligo with less than 1 year of follow up within the dataset.
* People over the age of 95 (for those reaching age 95 during the follow up period follow up was censored at age 95).
* People who have opted out of record sharing.

Max Age: 95 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Incident cases will be defined as people with a first ever diagnosis code of vitiligo during the study period. People with a diagnosis of vitiligo prior to the study period will be excluded. Each case will be assigned an index date at the time of their vitiligo diagnosis. Controls will be matched to people without Vitiligo matched on age, sex, ethnicity and deprivation.
Sampling Method: Non-Probability Sample
Enrollment: 39374 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2024-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew McGovern, MD, Study Director — Momentum Data
Locations (1):
- Momentum Data Limited, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data is confidential but can be made available in an anonymised form to bone fide researchers subject to the required data protection training and other requirements. All data will remain behind a firewall and will only be available for access through a secured computer network.
Supporting Information: SAP
Time Frame: There is no pre-specified time-frame for data availability; this will be considered on an individual basis for each request.
Access Criteria: As above.

REFERENCES:
- [Derived] Eleftheriadou V, Ahmed A, Nesnas J, Nagra R. The lifetime risk and impact of vitiligo across sociodemographic groups: a UK population-based cohort study. Br J Dermatol. 2024 Dec 23;192(1):63-71. doi: 10.1093/bjd/ljae282. PMID 39018020

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All adults and children (aged ≥ 13 years) contributing to the Optimum Patient Care Research Database (OPCRD) between 1 January 2004 and 31 December 2020, without a diagnosis of vitiligo prior to1 January 2004 were eligible for inclusion.
Pre-assignment Details: Participants with a diagnosis for an alternative depigmenting disorder or were diagnosed with vitiligo within 6 months of registering with their general practice (GP) were excluded.
Groups:
- People Without Vitiligo (Reference Group): Children and adults without Vitiligo registered with OPCRD during the study period
  No intervention: Observational analysis of usual care only.
Period: Overall Study
Arm/Group | People With Vitiligo | People Without Vitiligo (Reference Group)
Started | 7890 | 31484
Completed | 7890 | 31484
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- People With Vitiligo: Children (≥ 13 years) and adults with new onset Vitiligo registered with Optimum Patient Care Research Database during the study period.
  No intervention: Observational analysis of usual care only.
- People Without Vitiligo: Children (≥ 13 years) and adults without Vitiligo registered with Optimum Patient Care Research Database during the study period
  No intervention: Observational analysis of usual care only.
- Total: Total of all reporting groups
Arm/Group | People With Vitiligo | People Without Vitiligo | Total
Number analyzed (Participants) | 7890 | 31484 | 39374
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 43 [30 to 57] | 42 [30 to 59] | 42.5 [30 to 58]
Age, Customized [Count of Participants; unit: Participants]
  13-17 years | 487 | 1915 | 2402
  18-29 years | 1370 | 5471 | 6841
  30-49 years | 3063 | 12242 | 15305
  50+ years | 2970 | 11856 | 14826
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4131 | 16492 | 20623
  Male | 3759 | 14992 | 18751
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Ethnicity categorized according to the UK's Office for National Statistics definitions of major UK ethnic groups
  Participants
    White | 3726 | 14894 | 18620
    Black | 196 | 708 | 904
    Asian | 1197 | 4775 | 5972
    Mixed | 80 | 332 | 412
    Other | 299 | 1220 | 1519
    Not recorded | 2392 | 9555 | 11947
Index of Multiple Deprivation [Count of Participants; unit: Participants] — Index of Multiple Deprivation (IMD) is a UK national deprivation measure of deprivation which is based on the patient postcode. IMD has been stratified into quintiles with IMD 1 representing most deprived and IMD 5 being the least deprived.
  Participants
    1 (most deprived) | 1525 | 6094 | 7619
    2 | 1392 | 5545 | 6937
    3 | 1355 | 5418 | 6773
    4 | 1527 | 6084 | 7611
    5 (least deprived) | 1484 | 5928 | 7412
    Not recorded | 607 | 2415 | 3022
Body Mass Index, Categorical [Count of Participants; unit: Participants] — Body Mass Index (BMI) is a based on a participants height and weight.
  Participants
    < 18.5 (underweight) | 269 | 1054 | 1323
    18.5-25 (normal weight) | 2324 | 8504 | 10828
    25-30 (overweight) | 2386 | 8938 | 11324
    30-35 (class I obesity) | 1137 | 4410 | 5547
    35-40 (class II obesity) | 372 | 1654 | 2026
    > 40 (class III obesity) | 214 | 940 | 1154
    Not recorded | 1188 | 5984 | 7172
Smoking status, Categorical [Count of Participants; unit: Participants]
  Never smoked | 2709 | 10000 | 12709
  Current smoker | 1229 | 6114 | 7343
  Ex-smoker | 3642 | 13435 | 17077
  Not recorded | 310 | 1935 | 2245
Alcohol consumption, Categorical [Count of Participants; unit: Participants]
  None | 2605 | 10014 | 12619
  Within limits | 2913 | 11376 | 14289
  In excess of limits | 1005 | 3685 | 4690
  Harmful | 121 | 463 | 584
  Not recorded | 1246 | 5946 | 7192

OUTCOME MEASURES:

1. Primary Outcome: Risk of Depression Within Patients With Vitiligo
Description: Adjusted odds ratio calculated using logistic regression.
Time Frame: 2 years
Measure: Number; unit: Events
Groups:
- People With Vitiligo: Children (≥ 13 years) and adults with new onset Vitiligo
  No intervention: Observational analysis of usual care only.
- People Without Vitiligo: Children (≥ 13 years) and adults without Vitiligo (reference group)
  No intervention: Observational analysis of usual care only.
Arm/Group | People With Vitiligo | People Without Vitiligo
Number analyzed (Participants) | 7890 | 31484
Events | 1412 | 5395
Statistical Analysis 1: Comparison: People Without Vitiligo; Test type: Superiority; Odds Ratio (OR) = 1.08, 95% CI 2-sided [1.01 to 1.15] — Calculated as the odds of a person diagnosed with vitiligo having with depression versus people not diagnosed with vitiligo

2. Primary Outcome: Risk of Anxiety Within Patients With Vitiligo
Description: Adjusted odds ratio calculated using logistic regression.
Time Frame: 2 years
Measure: Number; unit: Events
Arm/Group | People With Vitiligo | People Without Vitiligo
Number analyzed (Participants) | 7890 | 31484
Events | 708 | 2430
Statistical Analysis 1: Comparison: People Without Vitiligo; Test type: Superiority; Odds Ratio (OR) = 1.19, 95% CI 2-sided [1.09 to 1.30] — Calculated as the odds of people diagnosed with vitiligo having anxiety compared to people not diagnosed with vitilligo

3. Primary Outcome: Risk of Depression or Anxiety Within Patients With Vitiligo
Description: Adjusted odds ratio of depression or anxiety in people with vitiligo calculated using logistic regression .
Time Frame: 2 years
Measure: Number; unit: Events
Arm/Group | People With Vitiligo | People Without Vitiligo
Number analyzed (Participants) | 7890 | 31484
Events | 1614 | 6064
Statistical Analysis 1: Comparison: People Without Vitiligo; Test type: Superiority; Odds Ratio (OR) = 1.10, 95% CI 2-sided [1.03 to 1.17] — Calculated as the odds of people diagnosed with vitiligo having anxiety or depression compared to people not diagnosed with vitilligo

4. Secondary Outcome: Primary Care Encounters
Description: Describe any disparities in primary care usage (primary care visits) reported as adjusted incidence rate ratios
Time Frame: 2 years
Measure: Number; unit: Events
Arm/Group | People With Vitiligo | People Without Vitiligo
Number analyzed (Participants) | 7890 | 31484
Events | 134207 | 439633
Statistical Analysis 1: Comparison: People Without Vitiligo; Test type: Superiority; Incidence rate ratio = 1.29, 95% CI 2-sided [1.26 to 1.32] — Adjusted incident rate ratio for increased primary care use was calculated by comparing patients with vitiligo versus matched controls not having vitiligo,using negative binomial regression

5. Secondary Outcome: Dermatology Referrals
Description: Percentage of participants diagnosed with vitligo and having a recorded dermatology referral event wthin two year estimated using using the Kaplan-Meier method.
Time Frame: 2 years
Population: Dermatology referrals were assessed only in patients with vitiligo
Measure: Number (95% Confidence Interval); unit: percentage of participants analyzed
Arm/Group | People With Vitiligo
Number analyzed (Participants) | 7890
percentage of participants analyzed | 20 [19 to 21]

6. Secondary Outcome: Mental Health Referrals
Description: Describe any disparities in healthcare utilisation ( mental health referrals) reported as adjusted hazard ratios
Time Frame: 2 years
Measure: Number; unit: Events
Arm/Group | People With Vitiligo | People Without Vitiligo
Number analyzed (Participants) | 7890 | 31484
Events | 311 | 1191
Statistical Analysis 1: Comparison: People Without Vitiligo; Test type: Other; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.93 to 1.20] — Hazard ratios for mental health referrals was calculated using Cox proportional hazards regression model and reflect a comparison of the incidence rates between people diagnosed with vitiligo and people not diagnosed with vitiligo

7. Secondary Outcome: Unemployment
Description: Describe any disparities in work-related impact (unemployment) reported as adjusted hazard ratios.
Time Frame: 2 years
Population: Subset of participants of working age
Measure: Number; unit: Events
Groups:
- People With Vitiligo: Adults aged 18-65 years with new onset Vitiligo
  No intervention: Observational analysis of usual care only.
- People Without Vitiligo: Adults aged 18-65 years without Vitiligo (reference group)
  No intervention: Observational analysis of usual care only.
Arm/Group | People With Vitiligo | People Without Vitiligo
Number analyzed (Participants) | 6241 | 23187
Events | 111 | 436
Statistical Analysis 1: Comparison: People Without Vitiligo; Test type: Other; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.76 to 1.15] — Hazard ratios for unemployment was calculated using Cox proportional hazards regression model and reflect a comparison of the incidence rates between people diagnosed with vitiligo and people not diagnosed with vitiligo

8. Secondary Outcome: Time Off Work
Description: Describe any disparities in work-related impact (time off work) reported as adjusted hazard ratios.
Time Frame: 2 years
Population: Subset of participants of working age
Measure: Number; unit: Events
Arm/Group | People With Vitiligo | People Without Vitiligo
Number analyzed (Participants) | 6241 | 23187
Events | 746 | 2472
Statistical Analysis 1: Comparison: People Without Vitiligo; Test type: Other; Hazard Ratio (HR) = 1.15, 95% CI 2-sided [1.06 to 1.24] — Hazard ratios for time off work was calculated using Cox proportional hazards regression model and reflect a comparison of the incidence rates between people diagnosed with vitiligo and people not diagnosed with vitiligo

9. Secondary Outcome: Sleep Disturbance
Description: Describe any disparities in sleep disturbance reported as adjusted hazard ratios.
Time Frame: 2 years
Measure: Number; unit: Events
Arm/Group | People With Vitiligo | People Without Vitiligo
Number analyzed (Participants) | 7890 | 31484
Events | 318 | 1102
Statistical Analysis 1: Comparison: People Without Vitiligo; Test type: Other; Hazard Ratio (HR) = 1.15, 95% CI 2-sided [1.02 to 1.31] — Hazard ratios for sleep disturbance was calculated using Cox proportional hazards regression model and reflect a comparison of the incidence rates between people diagnosed with vitiligo and people not diagnosed with vitiligo

ADVERSE EVENTS:
Description: Deaths, serious adverse events, and nonserious adverse events were not assessed for study participants.
Arm/Group | People With Vitiligo | People Without Vitiligo
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-25): https://cdn.clinicaltrials.gov/large-docs/94/NCT06097494/Prot_SAP_000.pdf